CLINICAL TRIAL: NCT05392569
Title: Intraoperative Evoked Potential Recording for Localization of Deep-Brain Stimulation Electrodes
Brief Title: Evoked Potential Recording During DBS Surgery
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Terence Sanger, Provost Associate Professor, University of Southern California
Other Study IDs: CCI-13-00324
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Movement Disorders in Children
MeSH Terms: interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Deep Brain Stimulation — In addition to standard micro electrode recordings, we propose to measure:
  1. surface potentials at the scalp (EEG) evoked by stimulation at the DBS electrode site
  2. micro electrode potentials at the DBS electrode site evoked by stimulation at the median and tibial nerves
  3. local field potentials at the DBS electrode site evoked by stimulation at the median and tibial nerves
  4. surface EMG in the first dorsal interosseus and gastrocnemius muscles during stimulation at the DBS electrode site.

SUMMARY:
Deep brain stimulation (DBS) has been approved for treatment of dystonia by the FDA under a humanitarian device exemption (HDE) status. DBS has been shown to be very effective in the treatment of a variety of diseases such as Parkinson's disease and essential tremor. It has been widely used for the treatment of primary and secondary dystonia as well. Surgery involves the placement of the DBS electrode in one or two of the deep nuclei constituting the basal ganglia. A subcutaneous thoracic or abdominal implantable pulse generator is placed and connected to the intracranial electrode. Pulsatile stimulation of the deep brain nuclei has been shown to result in significant improvement in many patients, including restoration of the ability to walk or make voluntary arm movements. A major difficulty with DBS is the accurate placement of the electrode. Adult patients are usually awakened during surgery and micro electrode recordings are used to determine the optimal electrode effectiveness and monitor for side effects. This requires the patient to be awake and cooperate, while on the operating table. When DBS is performed in children, such testing is often not possible because the children are scared or not cooperative when awakened during surgery, the procedure is most often done for Dystonia, which does not respond immediately, and dystonia may cause involuntary movements that could be dangerous in the operating room while the child's brain is exposed. As part of the routine clinical evaluation of target location in the operating room or Neuromodulation Unit, stimulation is performed using the deep brain or depth electrodes, typically at frequencies between 60hz and 185hz. For this research study, stimulation will occur at much lower frequencies, between 9hz and 20hz in order to be able to measure how electrical activity from the deep electrodes spreads to other electrodes or the scalp. As part of the research, peripheral nerves will also be stimulated at the wrist and knee at frequencies of 20hz to 150hz in order to measure the transmission of peripheral nerve stimulation to these areas of the brain. The investigators hope these additional studies will allow discovery for mechanisms that lead to movement disorders including dystonia, and that knowledge of these mechanisms will allow the investigators to develop new, safer, and more effective treatments in the future.

ELIGIBILITY:
Inclusion Criteria:

* - Subjects 5 years of age and/or older (including adults, ages 18+)
* Has chronic, intractable (drug refractory), generalized dystonia
* DBS surgery must be clinically indicated

Exclusion Criteria:

* Contraindication to neurosurgery and or a potentially reversible cause of dystonia that does not include surgery.

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Has plans to be implanted with a deep brain stimulator device. Although Medtronic's product information indicate that DBS is for individuals 7 years of age and older some DBS centers such as UCSF have implanted kids younger for off-label use. By including children 5 years of age into our study, we do not exclude children that may receive DBS off-label.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2013-11-13 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Assessment of Change in Dystonia using the Barry Albright Dystonia Scale | 1,3,6,12 months
  The Barry-Albright Dystonia Scale (BADS) is the most common outcome measure reported in intervention studies for children with dyskinetic cerebral palsy. Dystonia severity is rated on a 5-point (0 - 4), criterion based, ordinal scale for eight body regions (eyes, mouth, neck, trunk, left/right upper extremities and left/right lower extremities. The minimum score value is 0 (least severe) and the maximum score value is 32 (most severe).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hernandez-Martin E, Arguelles E, Zheng Y, Deshpande R, Sanger TD. High-fidelity transmission of high-frequency burst stimuli from peripheral nerve to thalamic nuclei in children with dystonia. Sci Rep. 2021 Apr 19;11(1):8498. doi: 10.1038/s41598-021-88114-w. PMID 33875779